CLINICAL TRIAL: NCT03035890
Title: Use of Response-Adapted Hypofractionated Radiation Therapy to Potentiate the Systemic Immune Response to Checkpoint Inhibitors in Non-Small Cell Lung Cancer
Brief Title: Hypofractionated Radiation Therapy to Improve Immunotherapy Response in Non-Small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: West Virginia Clinical and Translational Science Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WVU010516
Record Dates: First submitted 2017-01-23; First posted 2017-01-30 (Estimated); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Non Small Cell Lung Cancer Metastatic
Keywords: NSCLC; Lung Cancer; Non Small Cell Lung Cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Radiation; Radiation Dose Hypofractionation; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Radiation Therapy + Immunotherapy (Experimental): 3-5 fraction course of radiation therapy to target lesion concurrent with an immuno-therapeutic agent
  Interventions: Radiation: Radiation; Drug: Immuno-Therapeutic Agent

INTERVENTIONS:
Radiation: Radiation — Radiation therapy will be administered in 3 or 5 fractions over 3-10 days, at a recommended dose of 8-15 Gy per fraction for 3 total fractions (total dose 24-45 Gy) or 6-10 Gy per fraction for 5 total fractions (total dose 30-50 Gy)
  Other Names: Hypofractionated Radiation
Drug: Immuno-Therapeutic Agent — Immune checkpoint inhibitors that are FDA approved for use in patients with metastatic NSCLC will be acceptable for use concurrently with radiotherapy in this trial. The choice of agents will be at the treating medical oncologist's discretion, and include:
  * Nivolumab 240mg or 3 mg/kg once every 2 weeks (14 day cycle)
  * Pembrolizumab 200mg or 2 mg/kg once every 3 weeks (21 day cycle)
  * Atezolizumab 1200 mg once every 3 weeks (21 day cycle)
  These agents should be continued per standard of care until either disease progression or unacceptable toxicity.
  Other Names: Immunotherapy

SUMMARY:
This study includes the additional use of radiation therapy in combination immunotherapy in order to determine whether the radiation may improve the response of non-small cell lung cancer to immunotherapy and to monitor any side effects.

DETAILED DESCRIPTION:
Preclinical data suggest that radiation therapy may be uniquely suited to combine with immune checkpoint inhibitors, since radiation can disrupt a tumor's physical barriers to T-cell infiltration and augment antigen presentation, thus serving as an "in situ personalized vaccine" to activate the immune system and potentially enhance the systemic response.

The rationale for this study is to determine the safety and efficacy of combined immune checkpoint inhibitors and radiation therapy in metastatic non-small cell lung cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV metastatic Non Small Cell Lung Cancer
* Measurable disease of at least 1.5 cm in greatest dimension at least 2 non-irradiated sites (except for lymph nodes, in which the short-axis dimension must be at least 1.5cm). There must be at least 1 visceral organ metastasis outside of the brain.
* History of prior cytotoxic chemotherapy (with or without concomitant radiation therapy) with subsequent distant (metastatic) disease relapse, or progression of disease while on chemotherapy.
* Participant must be planned to receive (or actively receiving) standard of care checkpoint inhibitor immune therapy. For those patients actively receiving checkpoint inhibitor immune therapy the duration of immune therapy at the time of enrollment must be 4 months or less.
* Life expectancy greater than 3 months

Exclusion Criteria:

* Active autoimmune disease, primary immunodeficiency syndrome, HIV/AIDS, or hepatitis B or C
* Oral corticosteroid dependency
* Uncontrolled or untreated active brain metastases/CNS disease
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-01-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Shaikh, MD, Principal Investigator — West Virginia University
Locations (1):
- WVU Cancer Institute - Mary Babb Randolph Cancer Center, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiation Therapy + Immunotherapy: 3-5 fraction course of radiation therapy to target lesion concurrent with an immuno-therapeutic agent
  Radiation: Radiation therapy will be administered in 3 or 5 fractions over 3-10 days, at a recommended dose of 8-15 Gy per fraction for 3 total fractions (total dose 24-45 Gy) or 6-10 Gy per fraction for 5 total fractions (total dose 30-50 Gy)
  Immuno-Therapeutic Agent: Immune checkpoint inhibitors that are FDA approved for use in patients with metastatic NSCLC will be acceptable for use concurrently with radiotherapy in this trial. The choice of agents will be at the treating medical oncologist's discretion, and include:
  * Nivolumab 240mg or 3 mg/kg once every 2 weeks (14 day cycle)
  * Pembrolizumab 200mg or 2 mg/kg once every 3 weeks (21 day cycle)
  * Atezolizumab 1200 mg once every 3 weeks (21 day cycle)
  These agents should be continued per standard of care until either disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Radiation Therapy + Immunotherapy
Started | 35
Completed | 34
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy + Immunotherapy
Number analyzed (Participants) | 35
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [58.5 to 70.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Best Overall Response
Description: Time to Best Overall Response is measured in months from the start of treatment until the best response is achieved. Both RECIST v1.1 and irRC criteria will be used. RECIST Criteria: Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): ≥30% decrease in the sum of the diameters of target lesions. Stable Disease (SD): Neither sufficient shrinkage for PR nor sufficient increase for PD. Progressive Disease (PD): ≥20% increase in the sum of the diameters of target lesions or appearance of new lesions. irRC Criteria: Complete Response (irCR): Disappearance of all lesions in two consecutive observations ≥4 weeks apart. Partial Response (irPR): ≥50% decrease in tumor burden compared with baseline in two observations ≥4 weeks apart. Stable Disease (irSD): Neither sufficient decrease for irPR nor sufficient increase for irPD. Progressive Disease (irPD): ≥25% increase in tumor burden compared with nadir in two consecutive observations ≥4 weeks apart.
Time Frame: From the start of treatment until disease progression up to 2 years.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Radiation Therapy + Immunotherapy
Number analyzed (Participants) | 34
months | 14 [5.4 to 23.5]

2. Secondary Outcome: Time to Progression Free Survival
Description: The duration of time from start of treatment to time of progression or death, whichever occurs first. For those patients with a CR or PR, the reference for progressive disease is the smallest measurements recorded since the treatment started.
  RECIST version 1.1 will be used to assess the local response of irradiated lesions only, taking as reference the baseline largest diameter:
  Complete Response (CR) - Disappearance of the irradiated lesion Partial Response (PR) - > 30% decrease in the single largest diameter of the irradiated lesion Stable Disease (SD) - Neither sufficient decrease in diameter to qualify as PR nor sufficient increase in diameter to qualify as PD Progressive Disease (PD) - > 20% increase in the single largest diameter of the irradiated lesion. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm (0.5 cm).
Time Frame: From the start of treatment until the date of documented progression or death assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radiation Therapy + Immunotherapy
Number analyzed (Participants) | 35
Months | 6.9 [4.3 to 26]

3. Secondary Outcome: Overall Survival
Description: Amount of time from treatment until death, reported via follow up visit or phone call.
Time Frame: From the start of treatment until the date date of death, or the last follow up date on which the participant was reported alive, assessed up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation Therapy + Immunotherapy
Number analyzed (Participants) | 35
months | 15 [11 to 40]

ADVERSE EVENTS:
Time Frame: 2 years
Description: Adverse events were assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 during hospitalization, follow up or by chart review.
Arm/Group | Radiation Therapy + Immunotherapy
All-Cause Mortality (participants affected / at risk) | 4/35
Serious Adverse Events (participants affected / at risk) | 25/35
Other Adverse Events (participants affected / at risk) | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy + Immunotherapy (N=35)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Constrictive pericarditis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 3 (3)
Pericardial tamponade (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 5 (5)
Pain (General disorders) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 5 (5)
Sepsis (Infections and infestations) | 4 (4)
Skin infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 2 (2)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy + Immunotherapy (N=35)
Anemia (Blood and lymphatic system disorders) | 13 (13)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Constrictive pericarditis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 6 (6)
Pericardial tamponade (Cardiac disorders) | 2 (2)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 4 (4)
Hypothyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Bloating (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 5 (5)
Duodenal hemorrhage (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3)
Death NOS (General disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Fever (General disorders) | 2 (2)
General disorders and administration site conditions - Other, specify (General disorders) | 4 (4)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 8 (8)
Sepsis (Infections and infestations) | 6 (6)
Urinary tract infection (Infections and infestations) | 2 (2)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 1 (1)
GGT increased (Investigations) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 9 (9)
Weight loss (Investigations) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 7 (7)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 3 (3)
Vascular disorders - Other, specify (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT03035890/Prot_SAP_001.pdf
  • Informed Consent Form (2019-10-09): https://cdn.clinicaltrials.gov/large-docs/90/NCT03035890/ICF_002.pdf